CLINICAL TRIAL: NCT00958022
Title: Phase I/ II Trial of Carboplatin and Etoposide Plus LBH589 for Previously Untreated Extensive Stage Small Cell Lung Cancer
Brief Title: Carboplatin and Etoposide Plus LBH589 for Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on the tolerabilty challenges of the combination
Sponsor: Ahmad Tarhini (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Ahmad Tarhini, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-035
Record Dates: First submitted 2009-08-10; First posted 2009-08-13 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Panobinostat; Carboplatin; Etoposide; Podophyllotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LBH589 and carboplatin with etoposide (Experimental): The main goal during the Phase I portion of this research study is to find out the highest and safest dose of LBH589 that can be given in combination with carboplatin with etoposide in subjects with lung cancer without causing severe side effects. The main goal of the Phase II portion of this study is to find how lung cancer responds to the LBH589 in combination with carboplatin and etoposide.
  This study will also investigate how the body processes the combination of LBH589 and carboplatin with etoposide.
  Interventions: Drug: LBH589 and carboplatin with etoposide

INTERVENTIONS:
Drug: LBH589 and carboplatin with etoposide — LBH589 will be given in oral formulation starting at a dose of 10 mg (Dose Level 1) 3x/week (2 days apart, e.g. Mon, Wed, Fri), during 2 weeks out of 3-weekly dosing schedule. After establishing the MTD at a 2 out 3 weeks dosing schedule, a 3 out of 3 weeks dosing schedule will be tested at that dose. This schedule will be adopted in the absence of limiting toxicities. Will be continued weekly after completion of 6 cycles of combo chemotherapy until progression or intolerable toxicities.
  Etoposide: Cycles 1-6: 100 mg/m² IV over 60 mins, Days 1-3 every 21 days for 6 cycles Carboplatin: commercially available as a sterile lyophilized powder available in single dose vials containing 50mg, 150mg, or 450mg of carboplatin. Each vial contains equal parts by weight of carboplatin & mannitol. Commercial supplies will be used for this study. It will be administered as an i.v. infusion over 30 minutes. The dose will be calculated based on patient's body weight at each treatment visit.
  Other Names: Etoposide: VP-16, VePesid, VP-16-213, EPEG, epipodophyllotoxin, NSC #141540; Carboplatin: Paraplatin, CBDCA, Paraplatin NovaPlus

SUMMARY:
The subjects are being asked to take part in the Phase I or Phase II portion of a research study of a new investigational drug, LBH589, in combination with chemotherapeutic agents, carboplatin with etoposide. LBH589 (made by Novartis Pharmaceuticals Corp.) is considered "investigational" because it has not been approved for commercial use in the treatment of cancer by the U.S. Food and Drug Administration (FDA). Etoposide and carboplatin are chemotherapeutic agents approved by the FDA for the treatment of for small cell lung cancer.

LBH589 is a drug that may slow down the growth of cancer cells or kill cancer cells by blocking certain enzymes (proteins produced by cells). LBH589 has shown effects against cancer in laboratory studies and in studies using animals; however, it is not known if this medicine will show the same activity in humans. As of May 2006, approximately 100 patients have received treatment with either an intravenous or capsule form of LBH589. Only the capsule form of LBH589 will be used in this study.

The main goal during the Phase I portion of this research study is to find out the highest and safest dose of LBH589 that can be given in combination with carboplatin with etoposide in subjects with lung cancer without causing severe side effects. The main goal of the Phase II portion of this study is to find how the subject's lung cancer responds to the LBH589 in combination with carboplatin and etoposide at the highest and safest dose that was given in Phase I.

The subject may be enrolled in either Phase I or Phase II of the trial, depending on when they entered the study, but they will not be enrolled in both phases.

This study will also investigate how the subject's body processes the combination of LBH589 and carboplatin with etoposide. To determine this, the investigators will measure the amount of study drug in the subject's blood. This will be done with a series of blood tests, called pharmacokinetic (PK) tests. Pharmacokinetics is the study of how the study drug moves through the body. Other purposes of this study will be to sample the subject's genetic material (DNA/RNA) as well as to determine biomarkers in their blood. (For some cancers, biomarkers are a way to measure the extent of their disease or the effects of treatment.) These samples will also be stored for future studies.

DETAILED DESCRIPTION:
Treatment plan

* LBH589 will be given in oral formulation starting at a dose of 10 mg (Dose Level 1) three times per week (doses will be given at least 2 days apart, e.g. Monday, Wednesday, Friday), 2 out of 3 weeks dosing schedule.
* After establishing the MTD of LBH589 at a 2 out 3 weeks dosing schedule, a 3 out of 3 weeks dosing schedule will be tested at that dose, and this schedule will be adopted in the absence of limiting toxicities.
* Carboplatin will be given on day 1, every 21 days, and etoposide on days 1,2,3 every 21 days for up to 6 cycles. LBH589 will be continued weekly, three times-a-week, without interruption after completion of 6 cycles of combination chemotherapy until progression, or intolerable toxicities.

In the phase I part and for cycle 1 only, for the purpose of the PK studies LBH589 will start the week prior to the first carboplatin/etoposide cycle and PD studies will be performed (week -1).

Study design and sample size:

This is a phase I/II study. Phase I: 15-24 patients (estimated; Three to six patients will be enrolled at each dose level); Phase II: 39 patients.

ELIGIBILITY:
Inclusion criteria Note: subjects with screening labs outside of the normal institutional limits (WNL) definition may be allowed if determined by the treating physician and the PI that the deviation from the normal institutional limits is minor.

1. Patients with extensive stage SCLC who have not received prior chemotherapy

   For the phase I portion of the study only (and not for phase II), patients with progressive advanced or metastatic cancer (any histology) are allowed. These patients must have progressed on one or more standard therapies for the disease, or have disease which is known to be incurable and poorly responsive to available systemic therapies. Priority will be given in patients with neuroendocrine tumors, such as:
   1. Carcinoid
   2. Extrapulmonary small cell carcinoma
   3. Peripheral neuroepithelioma
   4. Merkel cell tumor
   5. Neuroblastoma
   6. Large cell neuroendocrine cancer
   7. Esthesioneuroblastoma and other neuroendocrine carcinomas of the head and neck 1.2 For the phase I portion of the study only (and not for phase II), patients are allowed to have prior chemotherapy except for Etoposide and LBH589.
2. Measurable disease (RECIST) (for phase II part only)
3. Patients may not have received prior HDACi therapy, including valproic acid, for the treatment of any medical condition.
4. ECOG Performance Status of ≤ 2 (see Appendix 4)
5. Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
6. Patients must meet the following laboratory criteria:

   * Hematology:

     * Absolute neutrophil count (ANC) ≥ 1500/mm³
     * Platelets ≥ 100,000/mm³
     * Hemoglobin ≥ 9 g/dL
   * Biochemistry:

     * Total Bilirubin within normal institutional limits.
     * AST/SGOT and ALT/SGPT ≤ 2.5 x upper limit of normal (ULN)
     * Renal: serum creatinine < 2 ULN
     * Total serum calcium (corrected for serum albumin) or ionized calcium WNL
     * If total serum calcium is elevated >ULN, confirm with ionized Calcium.
     * Serum potassium WNl WNL
     * Serum sodium WNL
     * Serum albumin WNL
     * Patients with any elevated Alkaline Phosphatase due to bone metastasis can be enrolled
7. Baseline MUGA or ECHO must demonstrate LVEF ≥ the lower limit of the institutional normal as interpreted by the reading cardiologist.
8. TSH and free T4 within normal limits (patients may be on thyroid hormone replacement)
9. Blood pressure of <140/90.
10. Patients must have fully recovered from the effects of any prior surgery or radiation therapy. A minimum time period of 3 weeks should elapse between the completion of extensive radiation therapy for recurrent/metastatic disease and enrollment in the study.
11. If patient has history of brain metastases, brain lesions should have been treated with surgery and/or radiation and be stable on repeat imaging.
12. No history of prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, unless there is a 3-year disease-free interval.
13. Patients should temporarily stop certain Nonsteroidal Anti-inflammatory Drug (NSAIDS) starting 5 days prior to protocol therapy, as described in 6.5.1.
14. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of study treatment and must be willing to use two methods of contraception one of them being a barrier method during the study and for 3 months after last study drug administration. Sexually active males and their female partners must agree to use an accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the study. Oral contraceptives are generally metabolized by CYP3A4. Since the potential of LBH589 to induce CYP3A4 is unknown, patients who are using oral contraceptives as a method of contraception, and are sexually active, should use another effective contraceptive method.
15. All patients must have given signed, informed consent prior to registration on study.

Exclusion criteria

1. Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
2. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
3. Impaired cardiac function including any one of the following:

   * Screening ECG with a QTc > 450 msec confirmed by treating physician investigator prior to enrollment to the study
   * Patients with congenital long QT syndrome
   * History of sustained ventricular tachycardia
   * Any history of ventricular fibrillation or torsades de pointes
   * Bradycardia defined as heart rate < 50 beats per minute. Patients with a pacemaker and heart rate ≥ 50 beats per minute are eligible.
   * Patients with a myocardial infarction or unstable angina within 6 months of study entry
   * Congestive heart failure (NY Heart Association class III or IV)
   * Right bundle branch block and left anterior hemiblock (bifascicular block)
4. Uncontrolled hypertension. Patients with history of hypertension must be well-controlled (≤140/90) on a stable regimen of anti-hypertensive therapy.
5. Concomitant use of drugs with a risk of causing torsades de pointes (See Appendix 1.-1)
6. Concomitant use of CYP3A4 inhibitors (See Appendix 1.-2)
7. Patients with unresolved diarrhea > CTCAE grade 1
8. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
9. Other concurrent severe and/or uncontrolled medical conditions
10. Patients who have received chemotherapy, any investigational drug or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
11. Concomitant use of any anti-cancer therapy or radiation therapy.
12. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of oral LBH589.
13. Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom
14. Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
15. Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
16. Patients with peripheral neuropathy ≥ CTCAE grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of Target Lesions | 18 weeks

SECONDARY OUTCOMES:
Evaluation of Best Overall Response | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad A Tarhini, MD, Principal Investigator — UPMC/UPCI
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States